CLINICAL TRIAL: NCT03412201
Title: Safety, Tolerability and Efficacy of Rapid Optimization, Helped by NT-proBNP testinG, of Heart Failure Therapies
Acronym: STRONG-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heart Initiative (Other)
Collaborators: Hôpitaux Universitaires Saint-Louis-Lariboisière (Unknown); Momentum Research, Inc. (Industry); Roche Diagnostics GmbH (Industry); INSERM UMR-942, Paris, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHF201701
Record Dates: First submitted 2018-01-12; First posted 2018-01-26 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: Disease management; Medication therapy management; Biomarkers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, parallel group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Follow-up and management of heart failure medications provided by the patient's general physician and/or cardiologist according to local medical standards
  Interventions: Other: Usual Care
- High Intensity Care (Experimental): Follow-up and management of heart failure medications provided by specialists at participating institutions. Doses of oral heart failure medications optimized within 2 weeks, provided clinical assessments and laboratory measures indicate that it is safe to increase doses.
  Interventions: Other: High Intensity Care

INTERVENTIONS:
Other: Usual Care — Follow-up and management of heart failure medications provided by the patient's general physician and/or cardiologist according to local medical standards
  Arms: Usual Care
Other: High Intensity Care — Follow-up and management of heart failure medications provided by specialists at participating institutions. Doses of oral heart failure medications optimized within 2 weeks, provided clinical assessments and laboratory measures indicate that it is safe to increase doses.
  Arms: High Intensity Care

SUMMARY:
STRONG-HF is a multicenter, randomized, parallel group study designed to evaluate the efficacy and safety of up-titration of standard oral heart failure medications during hospitalization for acute heart failure. Patients admitted for acute heart failure will be randomized within 2 days before discharge to either usual care or intensification of treatment with a beta-blocker, a renin-angiotensin system blocker, and a mineralocorticoid receptor blocker ("high intensity care" arm). In the "high intensity care" arm, patients' clinical signs and symptoms of heart failure will be assessed, and routine laboratory measures and biomarkers will be measured, at frequent post-discharge visits. When these measures indicate that it is safe to do so, the doses of the oral heart failure medications will be increased to optimal levels. Patients will be followed through 180 days from randomization. Patients assigned to the usual care group will be followed by their general physician and/or cardiologist according to local medical standards. Patients who were screened but did not meet eligibility criteria will be followed for 90-day outcome. Randomized patients will be contacted at 180 days to assess outcomes.

DETAILED DESCRIPTION:
STRONG-HF is a multicenter, randomized, parallel group study designed to evaluate the efficacy and safety of up-titration of standard of care medical therapy including beta-blockers; angiotensin converting enzyme inhibitors (ACEi), angiotensin receptor blocker (ARB) or angiotensin receptor neprolysin inhibitor (ARNi); and mineralocorticoid receptor antagonist (MRAs), on morbidity and mortality when initiated and up-titrated early during hospitalization for acute heart failure (AHF). Optimal safety conditions will allow physicians to introduce and/or continue oral HF therapies during this "vulnerable phase" in AHF patients. Patients admitted for AHF with clinical signs of congestion and elevated circulating N-terminal pro-B-type natriuretic peptide (NT-proBNP) and who are not treated with optimal doses of oral heart failure (HF) therapies within 2 days before hospital discharge for AHF and who are hemodynamically stable will be randomized in a 1:1 ratio to either usual care (named "usual care" arm) or intensification of treatment with beta-blockers, and ACEi (or ARB) or ARNi and a MRA (named "high intensity care" arm). In the latter arm, repeated assessments of clinical signs and symptoms of heart failure, routine clinical laboratory measures including potassium, sodium, and creatinine as well as NT-ProBNP will foster, encourage and ensure the safety of the optimization of oral heart failure therapies. AHF patients who were screened but did not meet inclusion criteria, including low circulating NT-proBNP at visit 2, will be followed for 90-day outcome. Randomized patients will be contacted at 180 days to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission within the 72 hours prior to Screening for acute heart failure with dyspnea at rest and pulmonary congestion on chest X-ray, and other signs and/or symptoms of heart failure such as edema and/or positive rales on auscultation.
2. All measures within 24 hours prior to Randomization of systolic blood pressure ≥ 100 mmHg, and of heart rate ≥ 60 bpm.
3. All measures within 24 hours prior to Randomization of serum potassium ≤ 5.0 mEq/L (mmol/L).
4. Biomarker criteria for persistent congestion:
5. At Screening, NT-proBNP > 2,500 pg/mL.
6. At the time of Randomization (within 2 days prior to discharge), NT-proBNP > 1,500 pg/mL (to ensure the persistence of congestion) that has decreased by more than 10% compared to Screening (to ensure the acuity of the index episode).
7. At 1 week prior to admission, at Screening, and at Visit 2 (just prior to Randomization) either (a) <= ½ the optimal dose of ACEi/ARB/ARNi (see Table) prescribed, no beta-blocker prescribed, and <= ½ the optimal dose of MRA prescribed or (b) no ACEi/ARB/ARNi prescribed, <= ½ the optimal dose of beta-blocker prescribed, and <= ½ the optimal dose of MRA prescribed.
8. Written informed consent to participate in the study.

Exclusion Criteria:

1. Age < 18 or > 85 years.
2. Clearly documented intolerance to high doses of beta-blockers.
3. Clearly documented intolerance to high doses of renin-angiotensin system (RAS) blockers (both ACEi and ARB).
4. Mechanical ventilation [not including continuous positive airway pressure (CPAP)/bilevel positive airway pressure (BIPAP)] in the 24 hours prior to Screening.
5. Significant pulmonary disease contributing substantially to the patients' dyspnea such as forced expiratory volume during the 1st second (FEV1)< 1 liter or need for chronic systemic or nonsystemic steroid therapy, or any kind of primary right heart failure such as primary pulmonary hypertension or recurrent pulmonary embolism.
6. Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy (CRT) device implantation within 3 months, or percutaneous transluminal coronary intervention (PTCI), within 1 month prior to Screening.
7. Index Event (admission for AHF) triggered primarily by a correctable etiology such as significant arrhythmia (e.g., sustained ventricular tachycardia, or atrial fibrillation/flutter with sustained ventricular response >130 beats per minute, or bradycardia with sustained ventricular arrhythmia <45 beats per minute), infection, severe anemia, acute coronary syndrome, pulmonary embolism, exacerbation of chronic obstructive pulmonary disease (COPD), planned admission for device implantation or severe non-adherence leading to very significant fluid accumulation prior to admission and brisk diuresis after admission. Troponin elevations without other evidence of an acute coronary syndrome are not an exclusion.
8. Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
9. History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
10. Sustained ventricular arrhythmia with syncopal episodes within the 3 months prior to screening that is untreated.
11. Presence at Screening of any hemodynamically significant valvular stenosis or regurgitation, except mitral or tricuspid regurgitation secondary to left ventricular dilatation, or the presence of any hemodynamically significant obstructive lesion of the left ventricular outflow tract.
12. Active infection at any time during the AHF hospitalization prior to Randomization based on abnormal temperature and elevated white blood cells (WBC) or need for intravenous antibiotics.
13. Stroke or transient ischemic attack (TIA) within the 3 months prior to Screening.
14. Primary liver disease considered to be life threatening.
15. Renal disease or estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 [as estimated by the simplified Modification of Diet in Renal Disease (MDRD) formula] at Screening or history of dialysis.
16. Psychiatric or neurological disorder, cirrhosis, or active malignancy leading to a life expectancy < 6 months.
17. Prior (defined as less than 30 days from screening) or current enrollment in a congestive heart failure (CHF) trial or participation in an investigational drug or device study within the 30 days prior to screening
18. Discharge for the AHF hospitalization anticipated to be > 14 days from admission, or to a long-term care facility. Randomization must occur within 12 days following admission and within 2 days prior to anticipated discharge.
19. Inability to comply with all study requirements, due to major co-morbidities, social or financial issues, or a history of noncompliance with medical regimens, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures
20. Pregnant or nursing (lactating) women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
180-day all-cause mortality or heart failure readmission | 180 days
  Cumulative risk of either readmission for heart failure or death at 180 days

SECONDARY OUTCOMES:
Change in quality of life | 90 days
  Change from baseline to 90 days in quality of life as measured using the EQ-5D visual analogue scale (VAS) which ranges from 0 to 100 with a higher score representing a better outcome. "EQ-5D" is the official name of a quality of life instrument developed by EuroQol.
180-day all-cause mortality | 180 days
  Cumulative risk of death at 180 days
90-day all-cause mortality or heart failure readmission | 90 days
  Cumulative risk of either readmission for heart failure or death at 90 days

OTHER OUTCOMES:
180-day cardiovascular death | 180 days
  Cumulative risk of death due to cardiovascular cause at 180 days
90-day cardiovascular death | 90 days
  Cumulative risk of death due to cardiovascular cause at 90 days
90-day all-cause mortality | 90 days
  Cumulative risk of death at 90 days
180-day heart failure readmission | 180 days
  Cumulative risk of readmission for heart failure at 180 days
90-day heart failure readmission | 90 days
  Cumulative risk of readmission for heart failure at 90 days
Finkelstein-Schoenfeld hierarchical composite | 90 days
  Hierarchical composite endpoint comprising death, heart failure readmissions, and EQ-VAS analyzed using Finkelstein-Schoenfeld methodology
Change in NT-proBNP | 90 days
  Change from baseline to 90 days in NT-proBNP on the log scale
Change in weight | 90 days
  Change from baseline to 90 days in weight in kg
Changes in signs and symptoms of congestion: NYHA class | 90 days
  Changes from baseline to 90 days in New York Heart Association (NYHA) class which ranges from 1 to 4 with a higher class representing a worse outcome
Changes in signs and symptoms of congestion: orthopnea | 90 days
  Changes from baseline to 90 days in orthopnea rated on a scale from 0 to 3 with a higher score representing a worse outcome
Changes in signs and symptoms of congestion: peripheral edema | 90 days
  Changes from baseline to 90 days in peripheral edema rated on a scale from 0 to 3 with a higher score representing a worse outcome
Changes in signs and symptoms of congestion: rales | 90 days
  Changes from baseline to 90 days in rales rated on a scale from 0 to 3 with a higher score representing a worse outcome
Changes in signs and symptoms of congestion: JVP | 90 days
  Changes from baseline to 90 days in jugular venous pulse (JVP) rated on a scale from 1 to 4 with a higher score representing a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD PhD FESC, Principal Investigator — Inserm UMRS 942; Hôpitaux Universitaires Saint-Louis-Lariboisière, University Paris Diderot
Locations (78):
- Argentina (11):
  - Sanatorio de la Canada, Villa María, Córdoba Province
  - Chutro Srl Clinic, Córdoba
  - Del Prado Private Clinic, Córdoba
  - San Roque Hospital, Córdoba
  - Rosario Cardiovascular Institute, Rosario
  - Rosario Clinical Research Institute - Delta, Rosario
  - Modelo Cardiology Center, San Miguel de Tucumán
  - Diagnostic and Treatment Medical Clinic SA, Santa Fe
  - Santa Rosa Hospital, Santa Rosa
  - San Martin SA Clinic, Venado Tuerto
  - Fusavim Privada SRL Clinic, Villa María
- Austria (6):
  - Internal Med. 1, St. Josef Hospital Braunau, Braunau am Inn
  - Clin. Dep. Internal Med 3, University Hospital St. Poelten, Sankt Pölten
  - 1. Med. Dep, Donauspital, Vienna
  - Cardiology Department at Hietzing Hospital with Neurological Center Rosenhugel, Vienna
  - Dep. Of Cardiology, Medical Univ. Vienna, Vienna
  - Internal Med., LKH Villach, Villach
- Colombia (4):
  - Cardiovascular Diagnostic Center, Cartagena, Departamento de Bolívar
  - CEQUIN Cardiomet Foundation, Armenia, Quindío Department
  - Cardiomet Pereira Clinical Research Center Foundation, Pereira, Risaralda Department
  - Santander Ophthalmological Foundation, Bucaramanga, Santander Department
- France (7):
  - Auxerre Hospital Center, Auxerre
  - University Hospital of Beziers, Béziers
  - Center Hospital Regional University of Tours Trousseu Hospital, Chambray-lès-Tours
  - University Hospital Henri Mondor, Creil
  - CHU Dijon Burgundy F. Mitterand, Dijon
  - Hôpitaux Universitaires Saint-Louis-Lariboisière, University Paris Diderot, Paris
  - Center Hospital of Toulon, Toulon
- Hungary (3):
  - Buda Hospital of the Hospitaller Order of Saint John of God, Budapest
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - St. Rafael Hospital in Zala County, Zalaegerszeg
- Israel (2):
  - Barzilay MC Ashkelon, Ashkelon
  - Asaf Harofe MC, Ẕerifin
- Mozambique (2):
  - Dept of Medicine Research unit, Maputo Central Hospital, Maputo
  - Mavalane Hospital, National Institute of Health, Maputo
- Nigeria (2):
  - Amino Kano Teaching Hospital, Kano
  - Murtala Muhammad Specialist Hospital, Kano
- Russia (21):
  - State Budget HealthCare Institution "First City clinical hospital named after E.E. Volosevich", Arkhangelsk
  - Regional budget Healthcare Institution "Cardiological dispensary", Ivanovo
  - Federal State Budget Educational Institution of Higher Education "Moscow State Medico-Dental University n.a. A.I. Evdokimov", under Ministry of Health of the Russian Federation, Moscow
  - Federal State Budget Educational Institution of Higher Education "Moscow State University n.a. M.V. Lomonosov", independent division Medical research Educational Centre, Moscow
  - Moscow City Hospital # 81, Moscow, Moscow
  - Moscow State Budget Healthcare Institution City clinical Hospital 52 of Moscow Healthcare Department, Moscow
  - Primary Healthcare Unit of the RF Ministry of Internal Affairs in Moscow, Moscow
  - Russian National Research Medical University n.a. N.I.Pirogov based at City Clinical hospital n.a. V.M.Buyanov DZM, Moscow
  - SBHI of Moscow City clinical hospital 64 of Moscow Healthcare department, Moscow
  - State Budget HealthCare Institution of Moscow "City clinical hospital 15 n.a. O.M. Filatov under Department of HealthCare of Moscow", Moscow
  - State Budget HealthCare Institution of Moscow "City clinical hospital 29 n.a. N.E. Bauman under Department of HealthCare of Moscow", Moscow
  - State Budget HealthCare Institution of Mosocw "City clinical hospital 51 under Department of HealthCare of Moscow", Moscow
  - Saint-Petersburg State Budget HealthCare Institution "City hospital 38 n.a. N.A. Semashko", Pushkin
  - Municipal Government-financed Institution of Healthcare "City Emergency Hospital" of Rostov-on-Don City, Rostov-on-Don
  - Federal State Budgetary Educational Institution of Higher Education "Ryazan State Medical University named after academician I.P. Pavlov", Ryazan
  - Federal State Budget Educational Institution of Higher Education "North-West state medical university n.a. I.I. Mechnikov under the Ministry of Health of the Russian Federation", Saint Petersburg
  - Saint Petersburg State Budget Healthcare Institution Pokrovskaya City Hospital, Saint Petersburg
  - Saint-Petersburg State Budget Healthcare Institution City Hospital 15, Saint Petersburg
  - State Budget Institution "Saint Petersburg state budget research institution of first aid named after I. I. Dzhanelidze", Saint Petersburg
  - State Budget HealthCare Institution of Vladimir Region "City Hospital 4 of Vladimir", Vladimir
  - State Institution of Healthcare of Yaroslavl Region "Clinical Hospital 8", Yaroslavl
- Slovakia (10):
  - National Institute of Cardio and Vascular Diseases, Bratislava
  - V. Internal Clinic, LFUK and UNB Bratislava, Bratislava
  - Internal Department, Hospital with Polyclinic Brezno, Brezno
  - Internal Department, Dolnooravian Hospital of Dr. L.N.Jege, Dolný Kubín
  - Internal Department, Hospital with Polyclinic Lucenec, Lučenec
  - First Internal Clinic, Faculty Hospital with Polyclinic Nove Zamky, Nové Zámky
  - Department of Internal Medicine Hospital Rimavska Sobota, Rimavská Sobota
  - Department of Internal Medicine UVN SNP-FN, Ružomberok
  - Internal Department, NsP Spisska Nova Ves, Spišská Nová Ves
  - Internal Department Hospital Arm General L. Svobodu Svidnik, Svidník
- South Africa (2):
  - Groote Schuur Hospital, Cape Town
  - Nelson Mandela Academic Hospital, Walter Sisulu University, Mthatha
- Tunisia (8):
  - Habib Bougatfa Hospital, Bizerte
  - Regional Hospital of Jendouba, Jendouba
  - Fattouma Bourguiba Hospital, Monastir
  - Hedi chaker Hospital, Sfax
  - Charles Nicolle Hospital, Tunis
  - Habib Thameur Hospital, Tunis
  - La Rabta Hospital, Tunis
  - Military Hospital, Tunis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang X, Davison B, Adamo M, Arrigo M, Biegus J, Chioncel O, Cohen Solal A, Cotter G, Edwards C, Kimmoun A, Lam CSP, Mebazaa A, Metra M, Novosadova M, Pang PS, Sliwa K, Takagi K, Voors AA, Ezekowitz JA. Guideline-Directed Medical Therapy Use in the STRONG-HF Trial. Circ Heart Fail. 2025 Sep;18(9):e012716. doi: 10.1161/CIRCHEARTFAILURE.124.012716. Epub 2025 Jul 3. PMID 40605744
- [Derived] Myhre PL, Grupper A, Mebazaa A, Davison B, Edwards C, Takagi K, Adamo M, Arrigo M, Barros M, Biegus J, Celutkiene J, Cerlinskaite-Bajore K, Chioncel O, Cohen-Solal A, Damasceno A, Deniau B, Diaz R, Filippatos G, Gayat E, Kimmoun A, Ter Maaten JM, Metra M, Novosadova M, Pagnesi M, Pang PS, Ponikowski P, Saidu H, Sliwa K, Tomasoni D, Voors A, Cotter G, Lam CSP. Changes in Liver Function Tests, Congestion, and Prognosis After Acute Heart Failure: The STRONG-HF Trial. JACC Adv. 2025 Mar;4(3):101607. doi: 10.1016/j.jacadv.2025.101607. Epub 2025 Feb 21. PMID 39983609
- [Derived] Farmakis D, Davison B, Fountoulaki K, Liori S, Chioncel O, Metra M, Celutkiene J, Cohen-Solal A, Damasceno A, Diaz R, Edwards C, Gayat E, Novosadova M, Bistola V, Pang PS, Ponikowski P, Saidu H, Sliwa K, Takagi K, Voors AA, Mebazaa A, Cotter G, Filippatos G. Rapid Uptitration of Guideline-Directed Medical Therapies in Acute Heart Failure With and Without Atrial Fibrillation. JACC Heart Fail. 2024 Nov;12(11):1845-1858. doi: 10.1016/j.jchf.2024.06.010. Epub 2024 Aug 14. PMID 39152986
- [Derived] Arrigo M, Davison B, Edwards C, Adamo M, Ambrosy AP, Barros M, Biegus J, Celutkiene J, Cerlinskaite-Bajore K, Chioncel O, Cohen-Solal A, Damasceno A, Diaz R, Filippatos G, Gayat E, Kimmoun A, Lam CSP, Metra M, Novosadova M, Pagnesi M, Pang PS, Ponikowski P, Saidu H, Sliwa K, Takagi K, Ter Maaten JM, Tomasoni D, Voors AA, Cotter G, Mebazaa A. Characteristics, treatment, and outcomes of early vs. late enrollees of the STRONG-HF trial. Am Heart J. 2024 Aug;274:119-129. doi: 10.1016/j.ahj.2024.04.019. Epub 2024 May 12. PMID 38740532
- [Derived] Ambrosy AP, Chang AJ, Davison B, Voors A, Cohen-Solal A, Damasceno A, Kimmoun A, Lam CSP, Edwards C, Tomasoni D, Gayat E, Filippatos G, Saidu H, Biegus J, Celutkiene J, Ter Maaten JM, Cerlinskaite-Bajore K, Sliwa K, Takagi K, Metra M, Novosadova M, Barros M, Adamo M, Pagnesi M, Arrigo M, Chioncel O, Diaz R, Pang PS, Ponikowski P, Cotter G, Mebazaa A. Titration of Medications After Acute Heart Failure Is Safe, Tolerated, and Effective Regardless of Risk. JACC Heart Fail. 2024 Sep;12(9):1566-1582. doi: 10.1016/j.jchf.2024.04.017. Epub 2024 May 12. PMID 38739123
- [Derived] Celutkiene J, Cerlinskaite-Bajore K, Cotter G, Edwards C, Adamo M, Arrigo M, Barros M, Biegus J, Chioncel O, Cohen-Solal A, Damasceno A, Diaz R, Filippatos G, Gayat E, Kimmoun A, Leopold V, Metra M, Novosadova M, Pagnesi M, Pang PS, Ponikowski P, Saidu H, Sliwa K, Takagi K, Ter Maaten JM, Tomasoni D, Lam CSP, Voors AA, Mebazaa A, Davison B. Impact of Rapid Up-Titration of Guideline-Directed Medical Therapies on Quality of Life: Insights From the STRONG-HF Trial. Circ Heart Fail. 2024 Apr;17(4):e011221. doi: 10.1161/CIRCHEARTFAILURE.123.011221. Epub 2024 Mar 6. PMID 38445950
- [Derived] Cotter G, Deniau B, Davison B, Edwards C, Adamo M, Arrigo M, Barros M, Biegus J, Celutkiene J, Cerlinskaite-Bajore K, Chioncel O, Cohen-Solal A, Damasceno A, Diaz R, Filippatos G, Gayat E, Kimmoun A, Lam CSP, Metra M, Novosadova M, Pang PS, Pagnesi M, Ponikowski P, Saidu H, Sliwa K, Takagi K, Ter Maaten JM, Tomasoni D, Voors A, Mebazaa A. Optimization of Evidence-Based Heart Failure Medications After an Acute Heart Failure Admission: A Secondary Analysis of the STRONG-HF Randomized Clinical Trial. JAMA Cardiol. 2024 Feb 1;9(2):114-124. doi: 10.1001/jamacardio.2023.4553. PMID 38150260
- [Derived] Pagnesi M, Metra M, Cohen-Solal A, Edwards C, Adamo M, Tomasoni D, Lam CSP, Chioncel O, Diaz R, Filippatos G, Ponikowski P, Sliwa K, Voors AA, Kimmoun A, Novosadova M, Takagi K, Barros M, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G, Mebazaa A, Davison B. Uptitrating Treatment After Heart Failure Hospitalization Across the Spectrum of Left Ventricular Ejection Fraction. J Am Coll Cardiol. 2023 Jun 6;81(22):2131-2144. doi: 10.1016/j.jacc.2023.03.426. PMID 37257948
- [Derived] Adamo M, Pagnesi M, Mebazaa A, Davison B, Edwards C, Tomasoni D, Arrigo M, Barros M, Biegus J, Celutkiene J, Cerlinskaite-Bajore K, Chioncel O, Cohen-Solal A, Damasceno A, Diaz R, Filippatos G, Gayat E, Kimmoun A, Lam CSP, Novosadova M, Pang PS, Ponikowski P, Saidu H, Sliwa K, Takagi K, Ter Maaten JM, Voors A, Cotter G, Metra M. NT-proBNP and high intensity care for acute heart failure: the STRONG-HF trial. Eur Heart J. 2023 Aug 14;44(31):2947-2962. doi: 10.1093/eurheartj/ehad335. PMID 37217188
- [Derived] Cerlinskaite-Bajore K, Lam CSP, Sliwa K, Adamo M, Ter Maaten JM, Leopold V, Mebazaa A, Davison B, Edwards C, Arrigo M, Barros M, Biegus J, Chioncel O, Cohen-Solal A, Damasceno A, Diaz R, Filippatos G, Gayat E, Kimmoun A, Metra M, Novosadova M, Pagnesi M, Pang PS, Ponikowski P, Saidu H, Takagi K, Tomasoni D, Voors AA, Cotter G, Celutkiene J. Sex-specific analysis of the rapid up-titration of guideline-directed medical therapies after a hospitalization for acute heart failure: Insights from the STRONG-HF trial. Eur J Heart Fail. 2023 Jul;25(7):1156-1165. doi: 10.1002/ejhf.2882. Epub 2023 Jun 1. PMID 37191154
- [Derived] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Derived] Cotter G, Davison B, Metra M, Sliwa K, Voors AA, Addad F, Celutkiene J, Chioncel O, Cohen Solal A, Diaz R, Damasceno A, Duengen HD, Filippatos G, Goncalvesova E, Merai I, Ponikowski P, Privalov D, Sani MU, Takagi K, Shogenov Z, Saidu H, Mebazaa A. Amended STRONG-HF study design. Eur J Heart Fail. 2021 Nov;23(11):1981-1982. doi: 10.1002/ejhf.2348. Epub 2021 Oct 4. No abstract available. PMID 34529313
- [Derived] Kimmoun A, Cotter G, Davison B, Takagi K, Addad F, Celutkiene J, Chioncel O, Solal AC, Diaz R, Damasceno A, Duengen HD, Filippatos G, Goncalvesova E, Merai I, Metra M, Ponikowski P, Privalov D, Sliwa K, Sani MU, Voors AA, Shogenov Z, Mebazaa A. Safety, Tolerability and efficacy of Rapid Optimization, helped by NT-proBNP and GDF-15, of Heart Failure therapies (STRONG-HF): rationale and design for a multicentre, randomized, parallel-group study. Eur J Heart Fail. 2019 Nov;21(11):1459-1467. doi: 10.1002/ejhf.1575. Epub 2019 Aug 19. PMID 31423712